CLINICAL TRIAL: NCT06949254
Title: PRospective Observational Study of STereotactic Body rAdiation Therapy With Androgen Deprivation Therapy for Organ-confined High-risk Prostate Cancer: the PROSTAR Trial
Acronym: PROSTAR
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: accord healthcare italia srl (Unknown)
Responsible Party: Sponsor
Other Study IDs: PROSTAR
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: High Risk Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples

GROUPS / COHORTS (1):
- high risk prostate cancer patient

SUMMARY:
Prostate Cancer (PCa) is the second most common malignancy and the 5th common cause of cancer-related mortality in men worldwide. The majority of patients with PCa is diagnosed with potentially curable disease and its management includes different approaches, such as surgery, Radiation Therapy (RT) and Androgen Deprivation Therapy (ADT), for exclusive use or in combination each other. Randomized clinical trials have shown that moderate hypofractionated RT (i.e., 2.5-4 Gy per fraction) has become a valid alternative to conventionally fractionated RT in patients with PCa. The rationale of hypofractionation is based on the strong radiobiological evidence of the low α/β ratio of PCa cells (1.5-2 Gy) and the greater sensitivity to high dose per fraction. Data suggests that prostate Stereotactic Body Radiation Therapy (SBRT) is an alternative treatment strategy for localized PCa with promising results in terms of disease control and toxicity, not inferior to conventionally fractionated RT. A systematic review of over 6000 men underwent prostate SBRT on prospective studies has demonstrated that this treatment provides favorable patient's quality of life, excellent disease control, and results in minimal serious acute or late toxicity.

Almost all the published studies, investigated the role of SBRT for organ-confined low- and intermediate favorable-risk disease. However, the HYPO-RT-PC trial addressed the role of SBRT in the context of unfavorable localized PCa. In this non-inferiority, phase III multicenter trial 1200 patients with either intermediate or high risk PCa were enrolled. The aim of the study was to demonstrate that SBRT (42.7 Gy in 7 fractions, 3 days per week, for 2.5 weeks) is non-inferior to conventional fractionation (78 Gy in 39 fractions, 5 days per week for 8 weeks) regarding failure-free survival, without significant differences in late normal tissues complications. Failure-free survival at 5 years was 84% in both treatment arms; adjusted HR was 1.002, hence ultra-hypofractionation was found to be non-inferior to conventional fractionated RT (given HR limit = 1.338). These results paved the way for the use of SBRT even in patients with unfavorable PCa. One controversial issue is the role of ADT in the setting of SBRT for localized PCa: in conventionally fractionated schedules, short term (4-6 months) and long term (1.5-3 years) ADT are considered the standard of care for unfavorable intermediate and high-risk PCa, respectively. However, in a systematic review/meta-analysis no benefit was found for ADT added to SBRT and similar results were reported also by King et al. in a retrospective study on over 1000 patients. The PACE C trial is one of three cohort of PACE that is multicenter, international phase 3 randomized controlled study. PACE C is set to explore the efficacy of SBRT in combination with ADT for patients with unfavorable intermediate and high-risk PCa and will recruit 1182 patients who will be randomized to receive either hypofractionated RT (60 Gy in 20 fractions) or SBRT delivered with 36.25 Gy in 5 fractions.

In this scenario, our study aims to evaluate the safety and efficacy of SBRT (40 Gy in 5 fractions every other day) coupled with ADT (relugolix 18-24 monthsaccording to clinical care) in patients with localized high-risk PCa.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ECOG performance status ≤ 2
* Histologically proven prostate adenocarcinoma
* High-risk group classification according to National Comprehensive Cancer Network (NCCN), defined by the presence of any one of the following high-risk factors: cT3-cT4 OR Grade Group 4 or Grade Group 5 OR PSA >20 ng/mL
* No pelvic nodal and distant metastases at staging with PSMA-PET
* IPSS ≤ 15 (alpha blockers allowed)
* Life expectancy of > 5 years
* Prostate volume ≤ 100 cc

Exclusion Criteria:

* Previous local radiation treatment of the prostate
* Previous radiotherapy to the pelvis
* Active Ulcerative Colitis or Crohn's Disease
* Previous tumors unless disease free for a minimum of 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients affected by localized high-risk prostate cancer candidate to radical radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of treatment efficacy: Biochemical-relapse free survival at 2 years (defined as rising PSA > 2 ng/mL above post-SBRT nadir). | from baseline to two years

SECONDARY OUTCOMES:
Biochemical-relapse free survival at 5 years (defined as rising PSA > 2 ng/mL above post-SBRT nadir) | from baseline to 5 years
Distant-metastases free survival at 2 years and 5 years | from baseline to 5 years
Cancer-specific survival at 2 and 5 years | from baseline to 5 years
Percentage analysis of ctDNA | from baseline to 5 years
  analysis of ctdna blood values at various timepoints to assess its concentration and evaluate the possible correlation with cancer and treatment. In particular calculation of the percentage of ctDNA over total cfDNA (Tumor Fraction percentage, TF%) at different timepoints.
  Evaluation of TF% variation in correlation with clinical parameters (e.g., disease progression) defined on the bases of the current clinical practice.
The role of ctDNA clearance as a biomarker to intercept the molecular relapse | from baseline to 5 years
  we want to assess ctdna clearance to see its possible correlation with a possible molecolar relapse, no unit of measure
EORTC QLQ-C30 for quality of life | from baseline to 5 years
  Questionnaire used to evaluate the general quality of life of patients, no score will be assessted
EORTC PR-25 questionnaires for the GU, GI and sexual domains at baseline and follow-up visits | from baseline to 5 years
  Questionnarie to assess the presence of possible side effects in the gastrointestinal tract, the questionnaire has no score.
International Prostatic Symptoms Score (IPSS) | from baseline to 5 years
  questionnaire used to evaluate the symptoms of prostatic hypertrophy. Minimum value = 0 (no symptoms), maximum value = 35 (severe symptomatology)
Urinary Incontinence (ICIQ-SF) | from baseline to 5 years
  questionnaire to evaluate urinary incontinence, minimum value = 0 (no urinary incontinence), maximum value = 19 (severe urinary incontinence)
International Index of Erectile Function 15 Item | from baseline to 5 years
  questionnarie to evaluate the erectile function. Minimum value = 0 (severe erectile disfunction), maximum value = 25 (normal sexual activity)
Serum PSA (ng/ml) at follow-up visits | from baseline to 5 years
Testosterone (ng/ml) levels at follow-up visits | from baseline to 5 years

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Humanitas Gavazzeni, Bergamo, Bergamo
  - Humanitas PIO X, Milan, Milan
  - IRCCS Humanitas Research Hospital, Rozzano, Milan